CLINICAL TRIAL: NCT05029466
Title: The Efficacy and Tolerability of Psilocybin in Participants With Treatment-Resistant Depression: a Phase 2, Randomized Feasibility Study
Brief Title: Psilocybin for Treatment-Resistant Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brain and Cognition Discovery Foundation (Other)
Collaborators: Braxia Scientific Corp. (Unknown); Usona Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 253490
Record Dates: First submitted 2021-08-20; First posted 2021-08-31 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Treatment Resistant Depression
Keywords: Bipolar II Disorder; Major Depressive Disorder; Depressive Disorder, Treatment-Resistant; Mood Disorders; Mental Disorders; Psilocybin; Hallucinogen; Psychedelic; Antidepressant; Phase 2; Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Bipolar Disorder; Depressive Disorder, Major; Mood Disorders; Mental Disorders; Depression | interventions — Psilocybin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment (Experimental): Participants will commence psilocybin treatment immediately upon study enrollment.
  Interventions: Drug: Psilocybin
- Delayed treatment (Experimental): Participants will commence psilocybin treatment two weeks after study enrollment.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a single dose of psilocybin and be assessed weekly for six weeks and biweekly for 18 weeks. Participants who relapse may receive up to two repeated doses of psilocybin.

SUMMARY:
The purpose of this study is to see if psilocybin, an investigational drug, is safe and well tolerated. Researchers also want to know if psilocybin can improve symptoms of depression. This study will see if psilocybin is safe and well tolerated by tracking changes in suicidal thoughts and behaviour, monitoring if any participants choose to stop participating in the study, and measuring any serious side effects, as well as how long they take to resolve. This study will also see if depression symptoms improve (or worsen) after psilocybin is administered. Additional information about participants' depressive symptoms and side effects will also be measured during the study.

DETAILED DESCRIPTION:
This randomized clinical trial will assess the feasibility, safety, and efficacy of single and repeat doses of psilocybin at point-of-care in persons with treatment-resistant depression as part of major depressive disorder or bipolar II disorder. The primary objective is to evaluate the feasibility of psilocybin in adults with treatment-resistant depression. The secondary objectives are to assess the efficacy and tolerability of psilocybin at point-of-care.

ELIGIBILITY:
Inclusion Criteria:

1. Over the age of 18 years and under the age of 65;
2. Diagnosed with major depressive disorder or bipolar II disorder by a healthcare provider;
3. Experiencing a major depressive episode (MDE) without psychotic features as defined and operationalized in the DSM-5, where the duration of the current episode is at least 3 months;
4. Have failed to respond to an adequate dose and duration of at least two guideline-concordant pharmacological treatments for the current MDE, as determined by the Massachusetts General Hospital-Antidepressant Treatment History Questionnaire; and
5. Able to complete all protocol required assessment tools without any assistance or alteration to the copyrighted assessments, and to comply with all study visits.

Individuals meeting one or more of the following DSM-5-defined criteria will be excluded:

* Current or past history of bipolar I disorder, schizophrenia, psychotic disorder, delusional disorder, paranoid personality disorder, or schizoaffective disorder, as assessed by a structured clinical interview (MINI) and International Personality Disorder Examination (IPDE);
* First degree history of schizophrenia or any psychotic disorders, including bipolar disorder with psychotic features;
* Currently experiencing symptoms of hypomania or mania as measured by the Young Mania Rating Scale (YMRS) total score > 12;
* History of a hypomanic or manic episode in the past 3 months;
* History of substance use and/or alcohol use disorder, of moderate severity or greater, in the past 3 months;
* Lifetime history of substance use disorder with a hallucinogen;
* Lifetime history of substance-induced psychosis;
* Currently experiencing psychotic symptoms as part of an MDE (mood congruent/mood incongruent).

Individuals meeting one or more of the following criteria will also be excluded:

* Exposure to psilocybin or any other psychedelic in the past 12 months prior to screening and/or during the current MDE;
* Uncontrolled or insulin-dependent diabetes;
* Seizure disorder;
* Other personal circumstances or behaviour judged to be incompatible with establishment of rapport or safe exposure to psilocybin;
* Women who are pregnant (self-report or via urine test), nursing, or planning a pregnancy;
* Refusal to use an effective contraceptive method by the participant or participant's partner (i.e., combined estrogen- and progestogen-containing hormonal contraception or progestogen-only hormonal contraception with inhibition of ovulation; intrauterine device; intrauterine hormone-releasing system; bilateral tubal occlusion; vasectomized partner; sexual abstinence) throughout their participation in the study;
* Recent stroke (< 1 year from signing of ICF), recent myocardial infarction (< 1 year from signing of ICF), uncontrolled hypertension (blood pressure > 140/90 mmHg) or clinically significant arrhythmia within 1 year of signing the ICF;
* Positive urine drug screen for illicit drugs or drugs of abuse at screening, a week prior to treatment, and during the trial (any positive urine drug test will be reviewed with participants to determine the pattern of use and eligibility will be determined at the investigator's discretion);
* Current enrolment in any investigational drug or device study or participation in such within 30 days of screening;
* Current enrolment in an interventional study for depression or participation in such within 30 days of screening;
* Abnormal and clinically significant results on the physical examination, vital signs, ECG, or laboratory tests at screening;
* Any other clinically significant cardiovascular, pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-19 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-22 (Actual)

PRIMARY OUTCOMES:
Feasibility of the study based on participant retention | Up to 24 weeks
  Participant drop-out rates will be calculated to determine the feasibility of psilocybin in adults with treatment-resistant depression.
Feasibility of the study based on suicidal ideation and behaviour scores | Up to 24 weeks
  Feasibility will be judged based on change in Columbia Suicide Severity Rating Scale (CSSRS) scores. The CSSRS evaluates suicidal ideation and behaviour. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).
Feasibility of the study based on adverse events | Up to 24 weeks
  Feasibility will be judged based on the percentage of participants experiencing serious adverse events and the percentage of adverse events resolving within 48 hours of each dose administration.

SECONDARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) total score | Up to 24 weeks
  The MADRS is a clinician-rated scale measuring depression severity, consisting of 10 items, each scored from 0 (normal) to 6 (severe), for a total possible score of 60; higher scores denote greater severity.
Montgomery-Åsberg Depression Rating Scale (MADRS) response rate | Up to 24 weeks
  The proportion of participants with at least a 50% reduction in MADRS total score relative to baseline.
Montgomery-Åsberg Depression Rating Scale (MADRS) remission rate | Up to 24 weeks
  The proportion of participants with a MADRS total score of 10 or lower.
McIntyre and Rosenblat Rapid Response Scale (MARRRS) | Up to 24 weeks
  The MARRS was recently validated in adults with treatment-resistant major depressive or bipolar disorder receiving open-label intravenous ketamine at a community-based treatment center The MARRRS is a self-reported 14-item self-report measure of depressive symptoms present during the past 72 hours. Total score ranges from 0 to 42; a higher score indicates greater symptom severity.
Patient Health Questionnaire 9-item (PHQ-9) | Up to 24 weeks
  The PHQ-9 is a self-rated measure of depressive symptom severity in the past two weeks. Each of the nine items is rated on a Likert scale, ranging from 0 (not at all) to 3 (nearly every day), and summed for a total score between 0 (no symptoms) to 27 (most severe).
Clinical Global Impressions Scale (CGI) | Up to 24 weeks
  The CGI severity module assesses the severity of a person's depressive illness using a seven-point Likert scale, ranging from "Normal, not at all depressed" to "Among the most extremely depressed patients". The CGI improvement module evaluates the global improvement of a person's condition since their last visit on a seven-point Likert scale, ranging from "Very much improved" to "Very much worse".
Quick Inventory for Depressive Symptomatology, Self-Report, 16-item (QIDS-SR-16) | Up to 24 weeks
  The QIDS-SR-16 total score ranges from 0 to 27 with 0 representing no depression and 27 representing severe depression.
Columbia Suicide Severity Rating Scale (CSSRS) | Up to 24 weeks
  The CSSRS evaluates suicidal ideation and behaviour. The suicidal ideation score ranges from 0 (no ideation) to 5 (active suicidal ideation with specific plan and intent). Suicidal ideation intensity score ranges from 0 (no ideation) to 25 (most severe). The presence of suicidal behaviour is rated as a binary response; the lethality of actual attempts are rated on a scale of 0 (no or very minor physical damage) to 5 (death) and the potential lethality of actual attempts are rated on a scale of 0 (behaviour not likely to result in injury) to 2 (behaviour likely to result in death despite available medical care).
Clinician-Administered Dissociative States Scale (CADSS), 23-item | Up to 20 weeks
  Total scores on the 23-item CADSS range from 0 to 92; a higher score denotes greater dissociative symptom severity.
Clinician-Administered Dissociative States Scale (CADSS), 6-item | Up to 20 weeks
  Total scores on the 6-item CADSS range from 0 to 24; a score of 3 or greater denotes the presence of dissociation symptom severity.
Brief Psychiatric Rating Scale (BPRS) | Up to 20 weeks
  The BPRS rating scale has 18 items, each item rated on a severity scale of 1 (not present) to 7 (extremely severe). 0 is entered if the item is not assessed.
Young Mania Rating Scale (YMRS) | Up to 20 weeks
  Total scores range from 0 to 60, with higher scores indicative of greater symptom severity.
Mystical Experiences Questionnaire (MEQ) | Up to 20 weeks
  The MEQ consists of 30 items, each item rated on a Likert scale (0-None/not at all to 5-Extreme, more than any other time in my life). The MEQ total score is computed by taking the average response to all items.
Sheehan Disability Scale (SDS) | Up to 24 weeks
  The SDS total score ranges from 0 to 30 with 0 representing no impairment and 30 representing severe impairment. The last two items of the scale (Days Lost and Days Unproductive) range from 0 to 7 (higher number denotes greater impairment).
EuroQol-5D 5-Level (EQ-5D-5L) | Up to 24 weeks
  The EQ-5D-5L consists of 5 items; each item ranges from 1 (no problems) to 5 (extreme problems). A participant's self-rated health is recorded on a vertical visual analogue scale (range 100 to 0), where the endpoints are labelled 'The best health you can imagine' (100) and 'The worst health you can imagine' (0).
World Health Organization-5 Well-Being Index (WHO-5) | Up to 24 weeks
  The WHO-5 is a measure of overall well-being, rated on a scale of 0 to 25, with higher scores denoting higher quality of life.
World Productivity and Impairment Questionnaire (WPAI) | Up to 24 weeks
  The WPAI is a six-item self-administered rating scale measuring work absenteeism, presenteeism, and productivity loss and daily activity impairment. Individuals are asked to rate to what extent health problems affected their ability to do regular daily activities other than work at a job (0-No effect on daily activities to 10-Completely prevented me from doing my daily activities). Respondents who are currently employed are additionally asked to rate the number of hours missed from work due to health problems, the number of hours missed due to other reasons (e.g., vacation, time off to participate in this study), and the number of hours worked in the past seven days, as well as to what extent health problems affected productivity while working (0-No effect on my work to 10-Completely prevented me from working). Responses to each question are scaled to an overall percentage score (0 to 100), with higher values denoting greater impairment
Perceived Deficits Questionnaire - Depression - 5-Item (PDQ-5-D) | Up to 24 weeks
  The total score ranges from 0 to 20, with greater scores indicative of greater subjective cognitive impairment.
Digit Symbol Substitution Test (DSST) | Up to 24 weeks
  The DSST assesses relative contributions of speed, memory, executive function and visual scanning. Participants are required to copy symbols that are paired with simple geometric shapes or numbers within 90 seconds for a total possible score of 0 to 90. A higher score reflects greater performance.
Trail Making Test A (TMT-A) | Up to 24 weeks
  The TMT is a two-part cognitive test. TMT-A assesses cognitive processing speed and consists of 25 circles distributed over a sheet of paper. Participants are asked to connect circles in numerical sequence. If a participant makes a mistake, the administrator points out the error, and the participant must return to the last correct circle and continue the task. Lower scores represent better performance.
Trail Making Test B (TMT-B) | Up to 24 weeks
  The TMT is a two-part cognitive test. TMT-B assesses executive functioning and consists of 25 circles distributed over a sheet of paper. Participants are asked to connect circles in alternating numerical and alphabetical sequence (e.g., 1-A-2-B). If a participant makes a mistake, the administrator points out the error, and the participant must return to the last correct circle and continue the task. Lower scores represent better performance.
Generalized Anxiety Disorder-7 (GAD-7) | Up to 24 weeks
  Total score ranges from 0 to 21; a higher score denotes greater symptom severity.
Snaith-Hamilton Pleasure Scale (SHAPS) | Up to 24 weeks
  The SHAPS total score ranges from 14 to 56, wherein a higher score indicates greater hedonic capacity (lower anhedonic severity).
Peripheral inflammatory and metabolic biomarkers | Up to 2 weeks
  Inflammatory, neuroplasticity, and metabolic targets that are hypothesized to be relevant to the therpeutic mechanism of psilocybin in depression (e.g., interleukin-6, brain-derived neurotrophic factor, insulin, leptin).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Rosenblat, MD, MSc, Principal Investigator — Canadian Rapid Treatment Centre of Excellence
Locations (1):
- Canadian Rapid Treatment Centre of Excellence (CRTCE), Mississauga, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosenblat JD, Meshkat S, Doyle Z, Kaczmarek E, Brudner RM, Kratiuk K, Mansur RB, Schulz-Quach C, Sethi R, Abate A, Ali S, Bawks J, Blainey MG, Brietzke E, Cronin V, Danilewitz J, Dhawan S, Di Fonzo A, Di Fonzo M, Drzadzewski P, Dunlop W, Fiszter H, Gomes FA, Grewal S, Leon-Carlyle M, McCallum M, Mofidi N, Offman H, Riva-Cambrin J, Schmidt J, Smolkin M, Quinn JM, Zumrova A, Marlborough M, McIntyre RS. Psilocybin-assisted psychotherapy for treatment resistant depression: A randomized clinical trial evaluating repeated doses of psilocybin. Med. 2024 Mar 8;5(3):190-200.e5. doi: 10.1016/j.medj.2024.01.005. Epub 2024 Feb 14. PMID 38359838